CLINICAL TRIAL: NCT06174337
Title: Autonomous Navigating Telepresence Robot for Alleviating Loneliness and Engaging Nursing Home Residents With and Without Dementia
Brief Title: Robot for Alleviating Loneliness and Engaging Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: Northeastern University (Other)
Collaborators: Vigorous Mind, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1R43AG073004-01 (NIH)
Record Dates: First submitted 2023-12-04; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Nursing Home Resident
Keywords: Robot; Loneliness; Nursing Home

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Use of Video Connection with Family via Robot — A remote family member is able to connect via video with a nursing home resident.

SUMMARY:
Social isolation is an emerging critical challenge in the care of older adults. Nursing home residents engage for an average of just 12 minutes per day with an activity director, a situation further exacerbated by Covid-19. Social isolation has detrimental effects on health, evidenced by 48.7% of nursing home residents with an active depression diagnosis, and 61% have moderate or severe cognitive impairment. The ultimate goal of this project is to alleviate older adults loneliness and boredom and to improve their mood in an economically feasible and scalable way. The investigators will integrate the existing Vigorous Mind (VM) multidomain activities platform for older adults with an affordable autonomous navigating robot to remotely socialize with and engage long-term-care facility (Facility) residents diagnosed with Mild Cognitive Impairment (MCI) or early-stage Alzheimer s disease or related dementias (Residents). The VM web-based platform has been used for group activities in senior living facilities for eight years. A Resident s profile in VM automatically searches the web and presents their favorite music, reminiscence content, comedy, and personalized brain exercises. VM is secure and HIPAA compliant. A VM employee (VM Companion) with experience running activities in a long-term care facility will be introduced by the staff to a Resident as a new companion who will visit the Resident through the robot to keep them company. The temi robot can be instructed to go to room 312 and it will navigate its way to the room. The Resident will be notified that the VM Companion is arriving for a visit, and once in the room, the VM Companion will see and greet the Resident, and the Resident will see the VM Companion. Since the VM Companion has dashboard access to the Resident s background and interests via the VM profile, they will be able to meaningfully socialize and engage in relevant VM activities. The goal of this Phase I project is to test the feasibility of this idea and to collect preliminary data on its effect on loneliness and mood.

DETAILED DESCRIPTION:
Background:

Social isolation and loneliness are critical challenges in older adult care. Loneliness is associated with declines in both physical and mental health. Approximately 50% of older adults over the age of 80 years experience loneliness. Nursing home residents are at a greater risk of loneliness due to limited staffing and COVID-19 visiting restrictions in place. More socially active older adults experience less cognitive decline in old age and better overall functioning. The use of technology for social interaction may have a positive impact on the behavioral and psychological symptoms of Alzheimer's disease (AD) especially in early stages of the disease. Robots are currently used in very few senior living facilities and cognitive support and communication are among the most desired functions. By using an autonomous navigating telepresence robot, the intervention brings the technology to the resident and allows her/him to socialize and interact with a loved-one without the need for a caregiver. This intervention integrates the Vigorous Mind system with the temi autonomous navigating telepresence robot (Vigorous Mind Robot - "VMR").

Aims:

1. Develop web-based visit scheduler and integrate the VM platform with the temi robot
2. Test usability of the VMR with 10 Residents and family members
3. Pilot study of the feasibility of a VMR intervention with 40 Residents

Experimental Design:

Testing of the VMR intervention consisted of a usability and feasibility phase. During usability, residents and family members were trained on use of the VMR robot and web-interface. Family members conducted two virtual visits and usability interviews with residents and family members followed each visit. Feasibility followed usability testing with a three-month period where family members were able to schedule virtual visits as often as they would like. Debriefing interviews with family members and residents occurred at the end of feasibility testing. Resident loneliness and mood was assessed with the UCLA Loneliness Scale, Geriatric Depression Scale, single-item loneliness scale, and PHQ-2.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years of age
* Able to read and speak English
* Recommended by staff or family member

Exclusion Criteria:

* Uncorrected vision or auditory impairment
* MoCA < 22

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Residents of 2 nursing homes in Massachusetts
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Overall experience with the robot - for the family | 3 months
  5 point Likert scale from maximum of "very good" to minimum of "very poor"
Overall experience with the robot for the resident | 3 months
  5 point Likert scale from maximum of "very good" to minimum of "very poor"
Ease of use of the robot for the family | 3 months
  5 point Likert scale from maximum of "very good" to minimum of "very poor"
Ease of use of the robot for the resident | 3 months
  5 point Likert scale from maximum of "very good" to minimum of "very poor"

SECONDARY OUTCOMES:
Change in Loneliness of resident | 3 months
  5 point rating from minimum of "seldom/never" to maximum of "always/often"; change over 3 months
Change in depression level of resident | 3 months
  Change in PHQ-2 score over 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New Bridge on the Charles, Dedham, Massachusetts
  - Maplewood Senior Living, Weston, Massachusetts

IPD SHARING:
Plan to Share IPD: No